CLINICAL TRIAL: NCT04194762
Title: Treadmill vs Cycling in Parkinson´s Disease Rehabilitation. Non-pharmacological, Randomized, Blind Rater, Clinical Trial for the Definition of the Most Effective Model in Gait Reeducation
Brief Title: PARK-FIT. Treadmill vs Cycling in Parkinson´s Disease. Definition of the Most Effective Model in Gait Reeducation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Sabela Novo Ponte, Principal Investigator, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.I.: 154/18
Record Dates: First submitted 2019-10-13; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: non pharmacological, randomised, double arm intervention. Treadmill training vs cycling training in equal intensity of exercise conditions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Intervention arm for each patient is masked for the raters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treadmill training (Experimental): Three training sessions per week for two months of treadmill. The intensity of exercise is monitored through the heart rate (HR). Patients ought to maintain a HR between 40 and 50% of the reserve HR
  Interventions: Other: Non pharmacological therapy
- Cycling (Active Comparator): Three training sessions per week for two months of cycling. The intensity of exercise is monitored through the heart rate (HR). Patients ought to maintain a HR between 40 and 50% of the reserve HR
  Interventions: Other: Non pharmacological therapy

INTERVENTIONS:
Other: Non pharmacological therapy — treadmill training and cycling training in equal intensity exercise.

SUMMARY:
PARK-FIT Treadmill vs Cycling in Parkinson´s Disease Rehabilitation. Non-pharmacological Clinical Trial for the Definition of the Most Effective Model in Gait Reeducation.

DETAILED DESCRIPTION:
Treadmill vs Cycling in Parkinson´s Disease Rehabilitation. Non-pharmacological Clinical Trial for the Definition of the Most Effective Model in Gait Reeducation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with idiopathic Parkinson's disease according to criteria from the United Kingdom Parkinson's Disease Society Brain Bank (UK-PDSBB)
* H&Y less than or equal to 2
* Stable drug treatment in the six weeks prior to the start of training and during the study.
* Signature of informed consent.

Exclusion Criteria:

* Diagnosis of other neuro-degenerative disease
* Cardiovascular disease or other systemic condition that contraindicates the moderate physical exercise
* Need for ambulation support
* Frequent freezing of gait events.
* Mni- Mental State Examination (MMSE) <26

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in step length after treadmill training or cycling. | Ten months
  Highlight changes in the length of the step after training in treadmill or cycling in patients with Parkinson´s disease.
Changes in step length after treadmill training. Discussion of its specificity to Parkinson´s disease | Ten months
  A description of step length and cadence for different velocities of gait after treadmill training.

SECONDARY OUTCOMES:
Rating Scale for Gait Evaluation in Parkinson's disease ( RSGE- PD scale ) | Ten months
  Gait status through the RSGE-PD Scale before and after the intervention.

OTHER OUTCOMES:
Movement Disorders Society- Unified Parkinson´s Disease Rating Scale II. (MDS-UPDRS II) | Ten months
  Motor functional status through the MDS-UPDRS II Scale before and after the intervention.
MDS-UPDRS III | Ten months
  Motor examination status through the MDS UPDRS III Scale before and after the intervention
The 39-item Parkinson´s Disease Questionnaire (PDQ-39) | Ten months
  Quality of life through the PDQ 39 Scale before and after the intervention.,

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886